CLINICAL TRIAL: NCT01214707
Title: Heart Rate Changes During Normal Activity, Exercise, and Seizures in Subjects With Epilepsy
Status: Completed | Type: Observational
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E-31
Record Dates: First submitted 2010-10-01; First posted 2010-10-05 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Epilepsy
Keywords: Exercise/No active Treatment
MeSH Terms: conditions — Epilepsy | interventions — Exercise

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Exercise protocol: No arms are required for this study as all subjects complete the entire protocol
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise during EMU stay
  Other Names: Exercise during EMU stay. No treatment intervention.

SUMMARY:
Characterization of the cardiac response (ECG) preceding an epileptic seizure.

DETAILED DESCRIPTION:
Characterization of the cardiac response (ECG) to physiologic events and comparison to changes in heart rate that precede an epileptic seizure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a clinical diagnosis of epilepsy requiring additional evaluation in an epilepsy monitoring unit (EMU).
2. Patient likely requires an EMU evaluation for a period of at least 3 days.
3. In the opinion of the Principal Investigator, the Patient is likely to have 3 - 5 seizures during the EMU stay.
4. Patient is currently taking at least one antiepileptic medication.
5. Patients must be 18 years or older and may be of either sex and of any race.
6. Patient must be in good general health, fully ambulatory, and able to complete the physical aspects of testing requirements.
7. Patient must be willing and able to complete informed consent and HIPAA authorization.
8. Patient is diagnosed with epilepsy but may also experience pseudo seizures or psychogenic seizures.

Exclusion Criteria:

1. Patients with severe psychiatric disease that in the investigator's judgment would prevent the patient's successful completion of the study.
2. Patients experiencing status epileptic within the last 6 months.
3. Patients with cardiovascular, respiratory, neuromuscular or gait disorders that in the investigator's judgment would cause unnecessary risk.
4. Patients prescribed drugs specifically for a cardiac or autonomic disorder that in the investigator's opinion would affect heart rate response. Drugs with secondary cardiac or autonomic actions are allowed.
5. Patients with cardiovascular arrhythmias or cardiac disease that would preclude the ability to detect intrinsic changes in heart rate due to exercise, stress, or seizure. This would include but not be limited to chronic atrial fibrillation and permanent cardiac pacemaker implantation.
6. Patients currently dependent on alcohol or narcotic drugs as defined by DSM IV-R.
7. Patients with a history of only psychogenic seizures or pseudo seizures.
8. Women who are pregnant. Women of childbearing age must take a pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with epilepsy already scheduled for an EMU stay.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Heart Rate Changes during Normal Activity, Exercise, and Seizures in Subjects with Epilepsy | 3 to 5 days
  Characterization of the cardiac response (ECG) to physiologic events and comparison to changes in heart rate that precede an epileptic seizure.

CONTACTS AND LOCATIONS:
Overall Officials: David M Treiman, MD, Principal Investigator — Barrow Neurological Institute Phoenix AZ; Ivan Osorio, MD, Principal Investigator — KUMC Kansas City, Kansas
Locations (2):
- United States (2):
  - BNI, Phoenix, Arizona
  - KUMC, Kansas City, Kansas